CLINICAL TRIAL: NCT04551599
Title: A Two-Part, Open-Label Phase 1 Study to Evaluate the Effect of Food and Age on the Pharmacokinetics of Danicopan
Brief Title: A Study of the Effects of Food and Age on Danicopan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ACH471-016
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: Factor D Inhibitor; Complement; Danicopan; Pharmacokinetics; Food-effect; Age-effect
MeSH Terms: interventions — danicopan

STUDY DESIGN:
Intervention Model Description: This will be 2-part study. Part 1 will be a randomized, 2-sequence, 2-period crossover study, and Part 2 will be a 1-period study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Sequence 1 (Experimental): Healthy, young, adult participants will receive danicopan once each Period as follows:
  Period 1: Danicopan administered under fed conditions.
  Period 2: Danicopan administered under fasted conditions.
  There will be a washout period of at least 7 days between the dose of danicopan in Period 1 and the dose of danicopan in Period 2.
  Interventions: Drug: Danicopan
- Part 1: Sequence 2 (Experimental): Healthy, young, adult participants will receive danicopan once each Period as follows:
  Period 1: Danicopan administered under fasted conditions.
  Period 2: Danicopan administered under fed conditions.
  There will be a washout period of at least 7 days between the dose of danicopan in Period 1 and the dose of danicopan in Period 2.
  Interventions: Drug: Danicopan
- Part 2 (Experimental): Healthy, elderly, male participants will receive a single dose of danicopan under fed conditions.
  Interventions: Drug: Danicopan

INTERVENTIONS:
Drug: Danicopan — A single dose of danicopan (200 milligrams) will be administered orally.
  Other Names: ACH-0144471; ALXN2040

SUMMARY:
This will be an open-label, 2-part study. Part 1 will be a randomized, 2-sequence, 2-period crossover, food-effect study in healthy young adult participants. Part 2 will be a 1-period age-effect study in healthy elderly male participants.

DETAILED DESCRIPTION:
This will be an open-label, 2-part study. Part 1 will be a randomized, 2-sequence, 2-period crossover, food-effect study in healthy young adult participants. Part 2 will be a 1-period age-effect study in healthy elderly male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Young adult males or females, between 18 and 55 years of age (Part 1 only).
2. Elderly male participants aged ≥ 65 years of age at screening (Part 2 only).
3. Body mass index in the range of 18.0 to 32.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50.0 kg at screening.
4. No clinically significant history or presence of electrocardiogram findings at screening.
5. Non-sterile male participants must agree to abstinence or use a highly effective method of contraception.
6. Female participants of childbearing potential must either agree to abstinence or to use, with their male partner, a highly effective method of contraception (Part 1 only).

Exclusion Criteria:

1. Clinically significant laboratory abnormalities.
2. Pregnant or lactating (Part 1 only).
3. History of any medical or psychiatric condition or disease that might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
4. History or presence of drug or alcohol abuse within previous 2 years, current tobacco user, and positive drugs-of-abuse or alcohol screen at screening or Day -1 of Period 1.
5. History of meningococcal infection, or a first-degree relative with a history of meningococcal infection.
6. Body temperature ≥ 38.0°Celsius at screening or prior to (first) dosing in Period 1 or history of febrile illness, or other evidence of infection, within 14 days prior to (first) dosing.
7. History of procedures that could alter absorption or excretion of orally administered drugs.
8. A history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs.
9. Major surgery within previous 4 weeks.
10. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days before (first) dosing, whichever is longer.
11. Donation of whole blood from 3 months prior to (first) dosing or of plasma from 30 days before (first) dosing, receipt of blood products within 6 months prior to (first) dosing, or receipt of a vaccine within 30 days prior to (first) dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Area Under The Concentration Versus Time Curve From Time 0 To The Last Measurable Concentration (AUC0-t) Of Danicopan Under Both Fed And Fasted Conditions In Healthy Young Adults | Up to 72 hours postdose
Area Under The Concentration Versus Time Curve From Time 0 Extrapolated To Infinity (AUC0-inf) Of Danicopan Under Both Fed And Fasted Conditions In Healthy Young Adults | Up to 72 hours postdose
Maximum Observed Concentration (Cmax) Of Danicopan Under Both Fed And Fasted Conditions in Healthy Young Adults | Up to 72 hours postdose
Time To Maximum Observed Concentration (Tmax) Of Danicopan Under Both Fed And Fasted Conditions in Healthy Young Adults | Up to 72 hours postdose
AUC0-t Of Danicopan Under Fed Conditions In Healthy Elderly Males | Up to 72 hours postdose
AUC0-inf Of Danicopan Under Fed Conditions In Healthy Elderly Males | Up to 72 hours postdose
Cmax Of Danicopan Under Fed Conditions In Healthy Elderly Males | Up to 72 hours postdose
Tmax Of Danicopan Under Fed Conditions In Healthy Elderly Males | Up to 72 hours postdose

SECONDARY OUTCOMES:
Number Of Healthy Young Adults And Healthy Elderly Males With Treatment-emergent Adverse Events | Day 1 (postdose) through follow-up (10 [+/- 2] days after last study drug administration)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Tempe, Arizona, United States